CLINICAL TRIAL: NCT00636506
Title: A Multi-Center Study to Assess the AMS IPP 2005 Inflatable Penile Prosthesis Cylinders, Pump and Reservoir.
Brief Title: Evaluation of the 2005 AMS (American Medical System) IPP (Inflatable Penile Prosthesis)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMS052
Record Dates: First submitted 2008-03-11; First posted 2008-03-14 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-05

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; Impotence
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AMS 700 IPP 2005 Implant Group (Experimental): Male subjects 21 years of age and older who are implanted with an AMS 700 IPP with MS (Momentary Squeeze) pump for erectile dysfunction.
  Interventions: Device: AMS 700 IPP with MS Pump

INTERVENTIONS:
Device: AMS 700 IPP with MS Pump — AMS 700 Series Inflatable Penile Prosthesis with MS Pump
  Other Names: AMS IPP 2005

SUMMARY:
The purpose of this study is to evaluate modifications to the AMS 700 Series pump, cylinders, reservoir and rear tip extender design, their impact on ease of use for the patient, and ease of implantation for the physician.

DETAILED DESCRIPTION:
Erectile dysfunction, the inability to attain or sustain a penile erection sufficient to permit satisfactory sexual intercourse, affects an estimated ten to 30 million men in the United States. Erectile dysfunction can be caused by many organic abnormalities, including diabetes mellitus, hypertension, vascular disease, neurogenic disorders, and other chronic diseases. Erectile dysfunction can be effectively treated with a variety of methods, including the implantation of an inflatable penile prosthesis. A multi-center trial is to be conducted to assess the AMS IPP 2002 Inflatable Penile Prosthesis including handling during IPP implantation procedures and short-term follow-up experience of subjects. The study will collect pre-operative information comparing the pump operation using scrotal models of the current pump with the study pump, and baseline erectile function history. Surgical data will be collected to assess device design and procedure enhancements. Patient and physician assessment of study device function, ease of use, ease of training/learning, and adverse events will be gathered post-operatively.

ELIGIBILITY:
1. Inclusion Criteria

   To be eligible to participate in this study, male subjects must meet the following requirements:
   1. The subject has been diagnosed with erectile dysfunction and has made an informed decision to be implanted with the AMS IPP 2005 Inflatable Penile Prosthesis Cylinder, Pump, and Reservoir.
   2. The subject has not had a previous penile prosthesis.
   3. The subject is willing and able to give written valid Informed Consent.
   4. The subject's reading level is judged adequate for reading and understanding the Informed Consent, patient questionnaires, and other study material
   5. The subject is ≥ 21 years of age.
   6. The subject has no known sensitivity to rifampin, minocycline or other tetracyclines as indicated in the device labeling.
   7. The subject does not have systemic lupus erythematosus
   8. The subject has the manual dexterity or mental ability to operate the pump.
   9. The subject does not have active urogenital infection or active skin infection in region of surgery as indicated in the device labeling.
   10. The subject is willing and able to return for follow-up evaluations and questionnaire completion according to the study protocol.
   11. The subject is an acceptable risk for anesthesia and surgery.
2. Exclusion Criteria

   Subjects will not be eligible for entry into this study if they meet any of the following criteria:
   1. The subject's reading level is judged inadequate for reading and understanding the Informed Consent, patient questionnaires, and other study materials.
   2. The subject is not willing or able to give written valid Informed Consent
   3. The subject meets any of the following contraindications for InhibiZone™ use:

   i. known allergy to or sensitivity to rifampin, minocycline, or to tetracyclines.

   ii. diagnosed with systemic lupus erythematosus. d) The subject has a current Urinary Tract Infection (UTI), urogenital infection, or active skin infection in the region of surgery.

   e) The subject does not have the manual dexterity or mental ability to operate the pump.

   f) The subject has a compromised immune system. g) The subject refuses to, or is unable to, comply with the requirements of the protocol or return for follow-up visits.

   h) The subject has been diagnosed with severe fibrosis due to priapism.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2005-08; Primary Completion 2006-02 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L. Dean Knoll, MD, Principal Investigator — Medical Research Associates of Nasville; Gerard D Henry, MD, Principal Investigator — Regional Urology LLC; Daniel Culkin, MD, Principal Investigator — University of Oklahoma Health Science Center; Dana A Ohl, MD, Principal Investigator — University of Michigan; Juan Otheguy, MD, Principal Investigator — Advanced Research Institute; Ridwan Shabsigh, MD, Principal Investigator — New York Center for Human Sexuality; Steven K Wilson, MD, Principal Investigator — Institute for Urologic Excellence
Locations (7):
- United States (7):
  - Institute for Urologic Excellence, Indio, California
  - Advanced Research Institute, New Port Richey, Florida
  - Regional Urology, LLC, Shreveport, Louisiana
  - University of Michigan School of Medicine, Ann Arbor, Michigan
  - New York Center for Human Sexuality, Brooklyn, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Medical Research Associates of Nashville, Nashville, Tennessee

REFERENCES:
- [Result] Knoll LD, Henry G, Culkin D, Ohl DA, Otheguy J, Shabsigh R, Wilson SK, Delk Ii J. Physician and patient satisfaction with the new AMS 700 momentary squeeze inflatable penile prosthesis. J Sex Med. 2009 Jun;6(6):1773-1778. doi: 10.1111/j.1743-6109.2009.01251.x. Epub 2009 Mar 30. PMID 19473458

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 76 subjects enrolled; 6 withdrew consent prior to the procedure, and 1 had the procedure aborted. 69 subjects were implanted with the study device; of these, 60 completed the study, 8 were lost to follow-up, and 1 had their device explanted.
Groups:
- AMS 700 IPP 2005 Implant Group: Male subjects 21 years of age and older who are implanted with an AMS 700 IPP with MS pump for erectile dysfunction.
Period: Overall Study
Arm/Group | AMS 700 IPP 2005 Implant Group
Started | 76
Completed | 60
Not Completed | 16
Not completed — Lost to Follow-up | 8
Not completed — Explanted | 1
Not completed — Withdrawal by Subject | 6
Not completed — Procedure aborted | 1

BASELINE CHARACTERISTICS:
Groups:
- AMS 700 IPP 2005 Implant Group: Male subjects 21 years of age and older who choose to undergo an IPP implantation for erectile dysfunction.
Arm/Group | AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 76
Region of Enrollment [Number; unit: participants]
  United States | 76

OUTCOME MEASURES:

1. Primary Outcome: Ease of Locating the Inflation Pump Bulb
Description: Physicians were asked to observe patients manipulating the device and to answer the question: "Could the subject easily locate the inflation pump bulb?" The response options were: Yes, No, and Not Tested
Time Frame: 4-8 weeks
Population: All subjects who were implanted and attended the device activation visit at 4-8 weeks post-op
Measure: Number; unit: Participants who easily located pumpbulb
Groups:
- AMS 700 IPP 2005 Implant Group at 4-8 Weeks: Male subjects 21 years of age and older who choose to undergo an IPP implantation for erectile dysfunction and who attended the 4-8 week follow-up visit.
Arm/Group | AMS 700 IPP 2005 Implant Group at 4-8 Weeks
Number analyzed (Participants) | 66
Participants who easily located pumpbulb | 63

2. Primary Outcome: Ease of Pumping Device to Full Erection
Description: Physicians were asked, "Compared to current AMS 700 pumps, please rate the ease of the inflation relating to the downward orientation of the AMS IPP 2005 pump bulb". Response options were on a 5-point Likert scale - Much easier; Somewhat easier; Same; Somewhat harder; Much harder.
Time Frame: 4-8 weeks post-op
Population: Subjects who attended the 4-8 week activation visit
Measure: Number; unit: Participants
Arm/Group | AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 66
Participants
  Much Easier | 28
  Somewhat Easier | 19
  Same | 3
  Somewhat Harder | 16
  Harder | 0

3. Primary Outcome: Quality of Erection (Suitability for Intercourse)
Description: Physicians were asked: "After inflation, did the erection appear suitable for sexual intercourse?" Response options were: Yes, No, Not Assessed
Time Frame: 4-8 weeks, 3 months, 6 months
Population: Subjects who attended the 4-8 week activation visit.
Measure: Number; unit: participants who answered yes
Groups:
- AMS 700 IPP 2005 Implant Group at 4-8 Weeks Follow-up: Male subjects 21 years of age and older who are implanted with an AMS 700 IPP with MS pump for erectile dysfunction at 4-8 weeks follow-up.
- AMS 700 IPP 2005 Implant Group at 3 Months Follow-up: Male subjects 21 years of age and older who are implanted with an AMS 700 IPP with MS pump for erectile dysfunction at 3 months follow-up.
- AMS 700 IPP 2005 Implant Group at 6 Months Follow-up: Male subjects 21 years of age and older who are implanted with an AMS 700 IPP with MS pump for erectile dysfunction at 6 months follow-up.
Arm/Group | AMS 700 IPP 2005 Implant Group at 4-8 Weeks Follow-up | AMS 700 IPP 2005 Implant Group at 3 Months Follow-up | AMS 700 IPP 2005 Implant Group at 6 Months Follow-up
Number analyzed (Participants) | 66 | 61 | 60
participants who answered yes | 66 | 60 | 59

4. Primary Outcome: Subjective Force Required to Inflate Device
Description: At the 3 and 6 month visit, subjects were asked to assess the force required to initiate inflation of the device. Response options were "Reasonable" and "Too Much"
Time Frame: 3 months, 6 months
Population: Subjects who attended the 3 month and/or 6 month follow-up visit
Measure: Number; unit: Participants
Groups:
- AMS 700 IPP 2005 Implant Group at 3 Months Follow-up; AMS 700 IPP 2005 Implant Group at 6 Months Follow-up: Male subjects 21 years of age and older who are implanted with an AMS 700 IPP with MS pump for erectile dysfunction.
Arm/Group | AMS 700 IPP 2005 Implant Group at 3 Months Follow-up | AMS 700 IPP 2005 Implant Group at 6 Months Follow-up
Number analyzed (Participants) | 61 | 58
Participants
  Reasonable | 50 | 48
  Too much | 11 | 9
  Missing | 0 | 1

5. Primary Outcome: Ability to Inflate Device Using One Hand
Description: Subjects were asked if they were able to inflate the device using one hand. Response options were: Yes, No
Time Frame: 3 months, 6 months
Population: All subjects who attended the follow-up visits
Measure: Number; unit: Participants
Groups:
- AMS 700 IPP 2005 Implant Group at 3 Months: Male subjects 21 years of age and older who are implanted with an AMS 700 IPP with MS pump for erectile dysfunction and who attended the 3 month follow-up visit.
- AMS 700 IPP 2005 Implant Group at 6 Months: Male subjects 21 years of age and older who are implanted with an AMS 700 IPP with MS pump for erectile dysfunction and who attended the 6 month follow-up visit.
Arm/Group | AMS 700 IPP 2005 Implant Group at 3 Months | AMS 700 IPP 2005 Implant Group at 6 Months
Number analyzed (Participants) | 61 | 58
Participants
  Yes | 31 | 33
  No | 30 | 23
  Missing | 0 | 2

6. Primary Outcome: Ease of Training Patient to Inflate Device Compared to the AMS Tactile Pump
Description: Physicians were asked: "Please rate the ease of training the subject to use the new AMS IPP 2005 pump in comparison to the AMS tactile pump." Response options were: Much easier, Somewhat easier, Same, Somewhat harder, Much harder
Time Frame: 4-8 weeks follow-up
Population: All subjects who attended the 4-8 week activation visit
Measure: Number; unit: Participants
Arm/Group | AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 66
Participants
  Much easier | 36
  Somewhat easier | 11
  Same | 5
  Somewhat harder | 13
  Much harder | 1

7. Primary Outcome: Ease of Training Patient to Inflate Device Compared to the Standard AMS 700 Pump
Description: Physicians were asked: "Please rate the ease of training the subject to use the new AMS IPP 2005 pump in comparison to the standard AMS 700 pump." Response options were: Much easier, Somewhat easier, Same, Somewhat harder, Much harder
Time Frame: 4-8 week activation visit
Population: All subjects who attended the 4-8 week activation visit
Measure: Number; unit: Participants
Arm/Group | AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 66
Participants
  Much easier | 39
  Somewhat easier | 18
  Same | 4
  Somewhat harder | 4
  Much harder | 1

8. Primary Outcome: Time to Complete Inflation
Description: Physicians were asked: "How much time was required for the subject to inflate?" Response options were: 0-30 seconds, 30-60 seconds, 60-90 seconds, 90-120 seconds, 2-3 minutes, Over 3 minutes
Time Frame: 4-8 week activation visit
Population: All subjects who attended the 4-8 activation visit
Measure: Number; unit: Participants
Arm/Group | AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 66
Participants
  0-30 seconds | 17
  30-60 seconds | 23
  60-90 seconds | 12
  90-120 seconds | 4
  2-3 minutes | 2
  Over 3 minutes | 8

9. Primary Outcome: Ease of Locating the Deflation Block
Description: Physicians were asked: "Could the deflation button be easily located?" Response options were: Yes, No, and Not Tested
Time Frame: 4-8 week activation visit
Population: All subjects who attended the 4-8 week activation visit
Measure: Number; unit: Participants
Arm/Group | AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 66
Participants
  Yes | 65
  No | 1
  Not tested | 0

10. Primary Outcome: Subjective Force Required to Initiate Deflation
Description: Subjects were asked: "The force required to initiate deflation was..." The response options were: "Too Much" and "Reasonable amount".
Time Frame: 3 months, 6 months
Population: All subjects who attended the follow-up visit
Measure: Number; unit: Participants
Groups:
- AMS 700 IPP 2005 Implant Group at 3 Months Follow-up: Subjects implanted with the AMS 700 IPP 2005 who attended the 3 month follow-up visit
- AMS 700 IPP 2005 Implant Group at 6 Months Follow-up: Subjects implanted with the AMS 700 IPP 2005 who attended the 6 month follow-up visit
Arm/Group | AMS 700 IPP 2005 Implant Group at 3 Months Follow-up | AMS 700 IPP 2005 Implant Group at 6 Months Follow-up
Number analyzed (Participants) | 61 | 58
Participants
  Reasonable | 54 | 51
  Too Much | 6 | 6
  No response | 1 | 1

11. Primary Outcome: Ability to Deflate Cylinders by Pressing the Deflation Button for Only a Few Seconds
Description: Physicians were asked to assess: "How long did you have to hold the deflation button for the deflation to set in motion?" The response options were: 1-2 seconds; 3-4 seconds; 5-6 seconds; 7-8 seconds; 9-10 seconds; More than 10 seconds, specify seconds.
Time Frame: 3 months, 6 months
Population: Physician assessment of all subjects who attended the 3 month and/or 6 month follow-up visit.
Measure: Number; unit: Percentage of Participants
Groups:
- 3 Months - AMS 700 IPP 2005 Implant Group: Male subjects 21 years of age and older who are implanted with an AMS 700 IPP with MS pump for erectile dysfunction and who attended the 3 month follow-up visit.
- 6 Months - AMS 700 IPP 2005 Implant Group: Male subjects 21 years of age and older who are implanted with an AMS 700 IPP with MS pump for erectile dysfunction and who attended the 6 month follow-up visit.
Arm/Group | 3 Months - AMS 700 IPP 2005 Implant Group | 6 Months - AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 61 | 59
Percentage of Participants
  1-2 seconds | 18.0 | 16.9
  3-4 seconds | 45.9 | 61.0
  5-6 seconds | 26.2 | 20.3
  7-8 seconds | 9.8 | 1.7
  9-10 seconds | 0 | 0
  More than 10 seconds | 0 | 0

12. Primary Outcome: Time to Complete Deflation
Description: Physicians were asked to assess: "How much time did it take for the device to deflate?" The response options were: 5-6 seconds; 7-8 seconds; 9-10 seconds; 10-15 seconds; 15-20 seconds; 20-25 seconds; 25-30 seconds; 35-40 seconds; 40-45 seconds; 45-50 seconds; More than 50 seconds, specify # of seconds
Time Frame: 3 months, 6 months
Population: Physician assessment of all subjects who attended the 3 month and/or 6 month follow-up visit.
Measure: Number; unit: Percentage of participants
Groups:
- 3 Months - AMS 700 IPP 2005 Implant Group: Male subjects 21 years of age and older who are implanted with an AMS 700 IPP with MS pump for erectile dysfunction attending the 3 month visit.
- 6 Months - AMS 700 IPP 2005 Implant Group: Male subjects 21 years of age and older who are implanted with an AMS 700 IPP with MS pump for erectile dysfunction attending the 6 month visit.
Arm/Group | 3 Months - AMS 700 IPP 2005 Implant Group | 6 Months - AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 61 | 58
Percentage of participants
  5-6 seconds | 18.3 | 20.7
  7-8 seconds | 13.3 | 17.2
  9-10 seconds | 20.0 | 27.6
  10-15 seconds | 21.7 | 10.3
  15-20 seconds | 16.7 | 12.0
  20-25 seconds | 3.3 | 6.9
  25-30 seconds | 6.7 | 1.7
  30-35 seconds | 0.0 | 0.0
  35-40 seconds | 0.0 | 3.4
  40-45 seconds | 0.0 | 0.0
  45-50 seconds | 0.0 | 0.0
  More than 50 seconds | 0.0 | 0.0

13. Primary Outcome: Ability to Deflate Device With One Hand
Description: "Could the subject easily deflate the AMS IPP 2005 with one hand?" The response options were: Yes; No; and Not Tested.
Time Frame: 3 months, 6 months
Population: All subjects who attended the 3 month and/or 6 month follow-up visit.
Measure: Number; unit: % who selected response option
Arm/Group | 3 Months - AMS 700 IPP 2005 Implant Group | 6 Months - AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 61 | 58
% who selected response option
  Yes | 50.8 | 56.9
  No | 49.2 | 39.7
  Missing | 0.0 | 3.4

14. Primary Outcome: Level of Flaccidity Achieved
Description: Physicians were asked "How would you rate the flaccidity of the AMS IPP 2005 cylinders at full deflation?" Response options were: Excellent; Very good; Good; Fair; Poor.
Time Frame: 4-8 weeks
Population: All subjects who attended the 4-8 week follow-up visit
Measure: Number; unit: Percentage of participants
Arm/Group | AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 66
Percentage of participants
  Excellent | 53.0
  Very Good | 34.8
  Good | 12.1
  Fair | 0.0
  Poor | 0.0

15. Primary Outcome: Ease of Training Patient to Deflate Device
Description: Physicians were asked to assess: "Please rate the ease of training the subject to use the new AMS IPP 2005 pump in comparison to the AMS Tactile Pump." The response options were: Much easier; Somewhat easier; Same; Somewhat harder; Much harder
Time Frame: 4-8 weeks
Population: All subjects who attended the 4-8 follow-up visit.
Measure: Number; unit: Percentage of participants
Groups:
- AMS Tactile Pump; Standard AMS 700 Pump: Male subjects 21 years of age and older who are implanted with an AMS 700 IPP with MS pump for erectile dysfunction.
Arm/Group | AMS Tactile Pump | Standard AMS 700 Pump
Number analyzed (Participants) | 66 | 66
Percentage of participants
  Much Easier | 54.5 | 59.1
  Somewhat Easier | 16.7 | 27.3
  Same | 7.6 | 6.1
  Somewhat harder | 19.7 | 6.1
  Much harder | 1.5 | 1.5

16. Primary Outcome: Patient Satisfaction With Deflation Mechanism
Description: Subjects were asked to assess: "Satisfaction with softness of penis when prosthesis is flaccid." Response options were: Very satisfied; Moderately satisfied; Somewhat satisfied; Somewhat dissatisfied; Moderately dissatisfied; Very dissatisfied
Time Frame: 3 Months, 6 Months
Population: All subjects who attended the 3 month and/or 6 month follow-up visit.
Measure: Number; unit: Percentage of participants
Arm/Group | 3 Months - AMS 700 IPP 2005 Implant Group | 6 Months - AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 61 | 58
Percentage of participants
  Very satisified | 42.6 | 56.9
  Moderately satisfied | 24.6 | 20.7
  Somewhat satisified | 16.4 | 17.2
  Somewhat dissatisfied | 13.1 | 3.4
  Moderately dissatisfied | 3.3 | 0.0
  Very dissatisified | 0.0 | 1.7

17. Primary Outcome: Ease of Dilation With the Reduced Angle of the Input Tubing
Description: Physicians were asked: "As compared to other devices, did the angle of the input tubing make it easier to insert?" Response options were: Yes; No/No effect
Time Frame: Time of implant (surgery)
Population: Physician assessment of each subject at time of implant
Measure: Number; unit: Percentage of participants
Arm/Group | AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 69
Percentage of participants
  Yes | 56.5
  No/No Effect | 43.5

18. Primary Outcome: Ease of Cylinder Placement With the Enhanced Profile of the Proximal Tip
Description: Physicians were asked: "How would you rate the overall ease of proximal insertion of the AMS IPP 2005 cylinders?" Response options were: Very easy; Moderately easy; Neither easy nor difficult; Moderately difficult; Very difficult
Time Frame: For duration of surgery
Population: Physician assessment of each subject at time of implant
Measure: Number; unit: Percentage of participants
Arm/Group | AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 69
Percentage of participants
  Very easy | 56.5
  Moderately easy | 27.5
  Neither easy nor difficult | 15.9
  Moderately difficult | 0.0
  Very difficult | 0.0

19. Primary Outcome: Comparison With Other Devices for Ease of Placement
Description: Physicians were asked: "Compared to other cylinders you have used, how would you rate the ease of proximal insertion of the AMS IPP 2005 cylinders?" Response options were: Much easier; Slightly easier; Same; Somewhat more difficult; More difficult
Time Frame: For duration of surgery
Population: Physician assessment of each subject at time of implant
Measure: Number; unit: Percentage of participants
Arm/Group | AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 69
Percentage of participants
  Much easier | 27.5
  Slightly easier | 37.7
  Same | 33.3
  Somewhat more difficult | 1.4
  More difficult | 0.0

20. Primary Outcome: Rating of the Rigidity of the Cylinders
Description: Physicians were asked: "How would you rate the rigidity of the AMS IPP 2005 cylinders at full inflation?" Response options were: Excellent; Very good; Good; Fair; Poor
Time Frame: 4-8 weeks follow-up
Population: All subjects who attended the 4-8 week follow-up visit
Measure: Number; unit: Percentage of participants
Arm/Group | AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 66
Percentage of participants
  Excellent | 40.9
  Very good | 43.9
  Good | 15.2
  Fair | 0.0
  Poor | 0.0

21. Primary Outcome: Ease of Insertion of New Flare Design Reservoir
Description: Physicians were asked: "As compared to the current 700 reservoir, how would you rate the ease of insertion of the AMS IPP 2005 reservoir?" Response options were: Much easier; Somewhat easier; Same; Somewhat harder; Much harder
Time Frame: For duration of surgery
Measure: Number; unit: Percentage of participants
Arm/Group | AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 69
Percentage of participants
  Much easier | 1.4
  Somewhat easier | 13.0
  Same | 84.1
  Somewhat harder | 1.4
  Much harder | 0.0

22. Primary Outcome: Ability of New Flare Design to Remain in Place
Description: Physicians were asked: "As comparable to the previous AMS 700 reservoir, does the new flare design of the AMS IPP 2005 reservoir retain its position as implanted?" Response options were: Yes; No
Time Frame: For duration of surgery
Population: Physician assessment of each patient at time of implant
Measure: Number; unit: Percentage of participants
Arm/Group | AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 69
Percentage of participants
  % Yes | 100
  % No | 0

23. Primary Outcome: Ease Attaching the New Snap Design Rear Tip Extender (RTE) to the Proximal Tip of the Cylinder
Description: Physicians were asked to assess their satisfaction level with the new snap design rear tip extender. Answer options were: Very satisfied; Moderate satisfied; Neutral; Moderately dissatisfied; Very dissatisfied.
Time Frame: For duration of surgery
Population: Physician assessment of each patient at time of implant for whom they used the RTEs (rear tip extenders)
Measure: Number; unit: percentage of physician responses
Arm/Group | AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 66
percentage of physician responses
  % Very satisfied | 50.0
  % Moderately satisfied | 16.7
  % Neutral | 28.8
  % Moderately dissatisfied | 1.5
  % Very dissatisfied | 3.0

24. Primary Outcome: Comparison Rating of the New Rear Tip Extender Design to Previous Design
Description: Physicians were asked, "Compared to AMS 700 RTE and other stackable RTE configurations, how would you rate the AMS IPP 2005 RTE configuration?" Answer options were: No RTEs implanted; Much better; Somewhat better; Same; Somewhat worse; Much worse
Time Frame: For duration of surgery
Population: Physician assessment of each patient for whom they used RTEs at time of implant
Measure: Number; unit: percentage of physician responses
Groups:
- AMS 700 IPP 2005 Implant Group With RTEs: Male subjects 21 years of age and older who are implanted with an AMS 700 IPP with MS pump for erectile dysfunction for whom physicians used RTEs.
Arm/Group | AMS 700 IPP 2005 Implant Group With RTEs
Number analyzed (Participants) | 66
percentage of physician responses
  % Much better | 40.9
  % Somewhat better | 25.8
  % Same | 31.8
  % Somewhat worse | 1.5
  % Much worse | 0.0

25. Primary Outcome: Physician Evaluation of the Pre-threaded Suture Needle for Ease of Removing Sheath
Description: Physicians were asked, "Was it easy to remove the blue suture sheath and white needle holder?" Answer options were: Yes; No, please explain
Time Frame: For duration of surgery
Population: Physician assessment of each patient at time of implant
Measure: Number; unit: percentage of physician responses
Arm/Group | AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 69
percentage of physician responses
  % Yes | 88.4
  % No | 11.6

26. Primary Outcome: Physician Evaluation of the Pre-threaded Suture Needle for Ease of Loading Furlow Tool
Description: Physicians were asked to assess the overall design compared to the current non-threaded design. Answer options: Significantly better; Better; Same; Worse; Significantly worse
Time Frame: For duration of surgery
Population: Physician assessment of each patient at time of implant
Measure: Number; unit: percentage of physician responses
Arm/Group | AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 69
percentage of physician responses
  % Significantly Better | 1.4
  % Better | 37.7
  % Same | 46.4
  % Worse | 14.5
  Significantly worse | 0.0

27. Primary Outcome: Physician Evaluation of OR Device Preparation Time
Description: Physicians were asked if the design of the pre-threaded needle facilitated faster loading of the Furlow tool. Answer options were: Yes; No
Time Frame: For duration of surgery
Population: Physician assessment of each patient at time of implant
Measure: Number; unit: percentage of physician responses
Arm/Group | AMS 700 IPP 2005 Implant Group
Number analyzed (Participants) | 69
percentage of physician responses
  % Assessed as Faster | 53.6
  % Assessed as Not as Fast | 46.4

ADVERSE EVENTS:
Description: Adverse events are assessed at the time of implant and at each follow-up visit.
Arm/Group | AMS 700 IPP 2005 Implant Group
Serious Adverse Events (participants affected / at risk) | 6/69
Other Adverse Events (participants affected / at risk) | 25/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMS 700 IPP 2005 Implant Group (N=69)
Urogenital Edema and Pain (Reproductive system and breast disorders) | 1 (1)
Device extrusion/erosion (Reproductive system and breast disorders) | 1 (1)
Device Infection (Infections and infestations) | 1 (1)
Cylinder Erosion (Reproductive system and breast disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1) — Not related to study device.
Urethral Erosion (Reproductive system and breast disorders) | 1 (1) — Not related to study device. Due to infected AUS (Artificial Urinary Sphincter)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMS 700 IPP 2005 Implant Group (N=69)
Device Auto-Inflation (Surgical and medical procedures) | 7 (7)
Device Aneurysm (Reproductive system and breast disorders) | 1 (1)
Mechanical Malfunction (Reproductive system and breast disorders) | 2 (2)
Pain/Discomfort with Ejaculation (Reproductive system and breast disorders) | 1 (1)
Pain/Discomfort with Erections (Reproductive system and breast disorders) | 1 (1)
Penile Sensation Change (Reproductive system and breast disorders) | 1 (1)
Seroma (Surgical and medical procedures) | 1 (1)
Pain/soreness with inflation/cycling of device (General disorders) | 6 (6)
Other (General disorders) | 1 (1) — Treated with retraining on pump
Not Device Related, Not Serious (General disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No